CLINICAL TRIAL: NCT01820845
Title: Accuracy of Pleth Variability Index (PVI) in Predicting Response to Intravenous Fluid Load During Scoliosis Surgery in Children
Brief Title: Accuracy of Pleth Variability Index (PVI) in Children
Acronym: PVI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PVI2013
Record Dates: First submitted 2013-01-28; First posted 2013-03-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Scoliosis
Keywords: Plethysmographic Variability Index; Esophageal Doppler; Scoliosis; Children; Age < 18 years; Scheduled for Scoliosis Surgery
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort of children with scoliosis surgery

SUMMARY:
Plethysmographic Variability index is a simple index accurate in predicting fluid responsiveness.

The aim of this study was to investigate its accuracy in predicting fluid response to intravenous fluid challenge during scoliosis surgery in children.

DETAILED DESCRIPTION:
The goal of the present study is to assess the validity of PVI in predicting the response to a fluid challenge during scoliosis surgery in children.

During this observational non-interventional study, each fluid challenge will be monitored by esophageal Doppler and PVI (Massimo Radical 5).

Anesthesia, surgery and intraoperative fluid administration id standardized according to our clinical protocol.

An increase in indexed Stroke Volume (iSV) by more than 15 % will define the positive response to the fluid challenge.

Fluid challenges will be performed in the supine position and in the prone position.

Statistical analysis will performed using the Receiving Operator Characteristics (ROC) curve with determination of the gray-zone allowing an error tolerance of 10 %.

ELIGIBILITY:
Inclusion Criteria:

* Scoliosis surgery
* Age < 18 years

Exclusion Criteria:

* Heart or vascular Diseases
* Rectal abnormalities
* Kidney Failure
* Neuromuscular scoliosis

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children undergoing scoliosis surgery
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plethysmographic Variability before each fluid challenge and percentage of variation in Indexed Stroke Volume during each fluid challenge. | During the intraoperative period.
  Data will be used to assess the accuracy of Plethysmographic Variability Index in predicting fluid challenge.

SECONDARY OUTCOMES:
Indexed Stroke volume before each fluid challenge and percentage of variation in indexed Stroke volume during each fluid challenge. | During the intraoperative period
  Data will be used to assess the accuracy of indexed Stroke volume in predicting the response to fluid challenge.

OTHER OUTCOMES:
Heart rate, Arterial pressure (systolic, diastolic and mean), End tidal CO2 concentration, Tidal volume, respiratory frequency, Airway pressure, Sevoflurane or desflurane concentrations before and after each fluid challenge. | During the intraoperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Robert Debre University Hospital, Paris, Paris, France

REFERENCES:
- [Result] Feldman JM, Sussman E, Singh D, Friedman BJ. Is the pleth variability index a surrogate for pulse pressure variation in a pediatric population undergoing spine fusion? Paediatr Anaesth. 2012 Mar;22(3):250-5. doi: 10.1111/j.1460-9592.2011.03745.x. Epub 2011 Dec 6. PMID 22142032